

# VIL DU DELTA I VÅR STUDIE SLIK AT KAN VI FORSKE PÅ SØVNBEHANDLINGEN DU VIL FÅ?

## FORMÅLET MED PROSJEKTET OG HVORFOR DU BLIR SPURT

Vi ønsker å kartlegge hvordan vi behandler pasientene våre og om dere blir bedre av behandlingen vi gir. Effekten av behandlingen på sikt er godt kjent i litteraturen, men effekten forløpende under behandling og av de ulike elementene i en klinisk pasientgruppe er i liten grad undersøkt. Noe av det vi ønsker å finne ut er om alle pasientene må ha alle de ulike elementene i behandlingen eller om behandlingen med fordel kan forenkles. Alle pasienter som blir behandlet ved Søvnklinikken vår blir spurt om å delta.

#### HVA INNEBÆRER PROSJEKTET FOR DEG?

I denne studien gir vi ingen annen behandling eller oppfølging enn det vi gjør vanligvis. Det innebærer også at du ikke skal fylle ut ekstra spørreskjemaer eller lignende om du deltar. Alle som deltar får den behandlingen som er klinisk anbefalt. Studien innebærer at vi kun registrerer det vi tilbyr deg av behandling og hva slags behandlingsresultater du opplever underveis og ved avslutning. Vi kommer til å registrere hva du svarer på spørreskjemaer og dine søvndagbøker, samt hvilken behandling vi gir deg. Dette er opplysninger som vi alltid uansett registrerer i din journal.

#### MULIGE FORDELER OG ULEMPER

I og med at du mottar vanlig behandling, er det ingen ulemper for deg ved å delta. Spesielt vi vil understreke at det ikke krever mer tid eller arbeid fra din side. Fordelen er at du bidrar til å gi oss mer kunnskap om hvordan vi behandler pasientene våre på Søvnklinikken og hvilke behandlingsresultater våre pasienter har.

#### FRIVILLIG DELTAKELSE OG MULIGHET FOR Å TREKKE DITT SAMTYKKE

Det er frivillig å delta i prosjektet. Dersom du ønsker å delta, undertegner du samtykkeerklæringen på siste side. Du kan når som helst og uten å oppgi noen grunn trekke ditt samtykke. Dette vil ikke få konsekvenser for din videre behandling. Dersom du trekker deg fra prosjektet, kan du kreve å få slettet innsamlede opplysninger, med mindre opplysningene allerede er inngått i analyser eller brukt i vitenskapelige publikasjoner. Dersom du senere ønsker å trekke deg eller har spørsmål til prosjektet, kan du kontakte prosjektleder og overlege Knut Langsrud (epost: knut.langsrud@stolav.no, telefon: 73864500).

### HVA SKJER MED OPPLYSNINGENE OM DEG?

Opplysningene som registreres om deg skal kun brukes slik som beskrevet i hensikten med prosjektet. Du har rett til innsyn i hvilke opplysninger som er registrert om deg og rett til å få korrigert eventuelle feil i de opplysningene som er registrert. Du har også rett til å få innsyn i sikkerhetstiltakene ved behandling av opplysningene. Alle opplysningene vil bli behandlet uten navn og fødselsnummer eller andre direkte gjenkjennende opplysninger. En kode knytter deg til dine opplysninger gjennom en navneliste. Det er kun prosjektleder som har tilgang til denne listen. Opplysningene om deg vil bli anonymisert eller slettet senest fem år etter prosjektslutt. Studiedataene planlegges brukt til 31.12.2030. Eventuelle utvidelser i bruk og oppbevaringstid kan kun skje etter godkjenning fra REK og andre relevante myndigheter.



## GODKJENNINGER

Regional komité for medisinsk og helsefaglig forskningsetikk har gjort en forskningsetisk vurdering og godkjent prosjektet (søknads-id hos REK: 710756)

Etter ny personopplysningslov har behandlingsansvarlig St. Olavs hospital, avdeling Østmarka, og prosjektleder Knut Langsrud et selvstendig ansvar for å sikre at behandlingen av dine opplysninger har et lovlig grunnlag.

Du har rett til å klage på behandlingen av dine opplysninger til Datatilsynet.

## KONTAKTOPPLYSNINGER

Dersom du har spørsmål til prosjektet, opplever uønskede hendelser eller bivirkninger, eller ønsker å trekke deg fra deltakelse, kan du kontakte prosjektleder og overlege Knut Langsrud (epost: knut.langsrud@stolav.no, telefon: 73864500).

TA MED DETTE SKJEMAET TIL DIN FØRSTE TIME VED SØVNKLINIKKEN.

JEG SAMTYKKER TIL Å DELTA I PROSJEKTET OG TIL AT MINE PERSONOPPLYSNINGER OG MITT BIOLOGISKE MATERIALE BRUKES SLIK DET ER BESKREVET

| Sted og dato | Deltakers signatur |
|--------------|-------------------------------------|
| | Deltakers navn med trykte bokstaver |